CLINICAL TRIAL: NCT05687799
Title: The Relationship of Neutrophil/Lymphocyte Ratio With Fatigue, Sleep and Quality of Life in Parkinson's Patients
Brief Title: Fatigue, Sleep and Quality of Life in Parkinson's Patients
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Asli Celik, MSc. Lecturer, Nigde Omer Halisdemir University
Other Study IDs: 2022/108
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Quality of life; Neutrophil/Lymphocyte ratio; Quality of sleep; Fatigue
MeSH Terms: conditions — Parkinson Disease; Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parkinson's Disease (PD) is a neurodegenerative disease characterized by chronic and progressive loss of dopaminergic neurons in the substantia nigra (SN) pars compacta. Sleep disturbances and fatigue are very common problems in Parkinson's patients. He reported that the frequency of fatigue was 47% in patients with a disease duration of less than five years and 70% in patients with a disease duration of more than five years. Fatigue in PD has been found to be associated with decreased physical activity, decreased functionality, sleep disorders, gait disturbances, motor findings, autonomic findings, increased levodopa dose, and motor fluctuations. Motor and non-motor symptoms in Parkinson's patients affect the individual's ability to perform activities of daily living independently. Impairments in functional status lead to negative consequences on quality of life. PD affects the individual not only physically, but also psychologically and socially.The neutrophil/lymphocyte ratio is a marker of peripheral inflammation. The relationship of peripheral inflammation to quality of sleep, quality of life and fatigue in individuals is unclear. The aim of this study was to investigation fatigue, quality of sleep and quality of life, and the relationship between neutrophil/lymphocyte ratio in Parkinson's patients.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a neurodegenerative disease characterized by chronic and progressive loss of dopaminergic neurons in the substantia nigra (SN) pars compacta. Sleep disturbances and fatigue are very common problems in Parkinson's patients. He reported that the frequency of fatigue was 47% in patients with a disease duration of less than five years and 70% in patients with a disease duration of more than five years. Fatigue in PD has been found to be associated with decreased physical activity, decreased functionality, sleep disorders, gait disturbances, motor findings, autonomic findings, increased levodopa dose, and motor fluctuations. Motor and non-motor symptoms in Parkinson's patients affect the individual's ability to perform activities of daily living independently. Impairments in functional status lead to negative consequences on quality of life. PD affects the individual not only physically, but also psychologically and socially.The neutrophil/lymphocyte ratio is a marker of peripheral inflammation. The relationship of peripheral inflammation to quality of sleep, quality of life and fatigue in individuals is unclear. The aim of this study was to investigation fatigue, quality of sleep and quality of life, and the relationship between neutrophil/lymphocyte ratio in Parkinson's patients.The aim of this study was to investigation fatigue, quality of sleep and quality of life, and the relationship between neutrophil/lymphocyte ratio in Parkinson's patients. A total of 39 Parkinson's Disease age of older the 50 participate in the research.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with idiopathic Parkinson's disease
* Healthy individuals who do not have musculoskeletal disease or any neurological disease that may affect assessments
* Older than 50 years old
* Volunteer to participate in the study
* Grade 1-3 on the Modified Hoehn-Yahr Scale
* To have a score above 24 in the Standardized Mini Mental Test
* To have a hemogram follow-up in the last 1 month before the date of participation in the study.
* Being able to walk independently on flat ground

Exclusion Criteria:

* Having an additional or psychiatric disease other than Parkinson's disease
* Lack of cooperation
* Presence of orthopedic problems (such as fractures, osteoporosis, osteomyelitis)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients who applied to Nigde Omer Halisdemir University Training and Research Hospital Neurology Clinic will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease Quality of Life-8 | Baseline
  One question from each of the eight domains in Parkinson's Disease Quality of Life-39, which are activities of daily living, physical discomfort, cognition, communication, emotional well-being, mobility, social support and stigma, gives the total domain score.Each question is scored between 0-4 points and points are added up. The total score is then divided by the total possible score and given as a percentage point out of 100. The lower the score, the higher the quality of life.
Hemogram | Baseline
  The neutrophil/lymphocyte ratio is a marker of peripheral inflammation.
Parkinson's Fatigue Scale-16 | Baseline
  The scale is the only fatigue scale specific to PD developed by Brown et al. It examines the impact of fatigue on daily life and consists of 16 items designed to assess the physical effects of fatigue. The scale allows to measure the presence of fatigue (seven items) and its effect on daily function (nine items). The subjects are asked to respond to the statements about fatigue between 1 (strongly disagree) and 5 (strongly agree). The higher score, the worsen fatigue scale in participant.
The Parkinson's Disease Sleep Scale | Baseline
  Parkinson's Disease Sleep Scale consists of 15 questions to be answered by the patient. With this, the quality of sleep as a whole during the night, difficulty in starting and maintaining sleep, night restlessness, nocturnal psychosis, nocturia, nocturnal motor symptoms, restlessness of sleep and naps during the day can be evaluated. The test is done by giving a score between 0 (very severe complaints) and 10 (no complaints) for each question. The total score point is 150. Higher scores indicate better sleep quality.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | Baseline
  This scale was created to evaluate the motor performance, mental and mental status, and activities of daily living of Parkinson's patients. It also evaluates motor fluctuations, dyskinesias, and autonomic dysfunction. The scale was prepared as 4 parts and 42 items. When the extremities are evaluated separately, it increases up to 55 items. Items are rated from 0 (no symptoms or signs) to 4 (most severe symptoms and signs). The first part evaluates the non- motor features of the disease, such as thoughts, behaviors, and emotions. The second part consists of activities of daily living. In the third part, motor examination, in the fourth part, the complications of the treatment are given. It is used to evaluate the symptoms of the disease and the complications that develop due to treatment. In this scale, which consists of 4 parts, the scoring of each item is between 0-4 points. The increase in the total score reflects the increase in the severity of the symptoms.
Modified Hoehn and Yahr Scale | Baseline
  This staging scale was developed by Margaret Hoehn and Melvin Yahr (1967) for use in describing the stage of Parkinson's disease. According to the staging scale, the disease is handled in 8 stages. The lower the stage, the better of the stage Parkinson's disease.
  Stage 0: No signs of disease Stage 1: Unilateral disease Stage 1.5: Unilateral plus axial involvement. Stage 2: Bilateral disease, no balance disorder. Stage 2.5: Mild bilateral disease recovering on pull test. Stage 3: Mild to moderate bilateral disease and some postural instability, physically independent.
  Stage 4: Severe disability, able to stand and walk unaided. Stage 5: Unassisted wheelchair or bed dependent.

OTHER OUTCOMES:
Standardized Mini Mental Test | Baseline
  There are 19 items in this test, which consists of 5 main parts: orientation, recording memory, attention and calculation, recall and language. The total score of the test is evaluated out of 30 and 24 points are accepted as the threshold value for the diagnosis of mild dementia. The higher the score, the higher the cognition of individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek İŞCAN, Dr., Principal Investigator — Nigde Omer Halisdemir University Treaning and Research Hospital
Locations (1):
- Nigde Omer Halisdemir University Treaning and Research Hospital, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No